CLINICAL TRIAL: NCT02403843
Title: RNS® System Post-Approval Study in Epilepsy
Brief Title: RNS® System Epilepsy Post-Approval Study
Acronym: PAS
Status: Active, not recruiting | Type: Observational
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Other Study IDs: NP10012; PMA100026 (Other: United States FDA)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Evaluation: A group of subjects with the RNS System implanted who elect to continue to receive RNS System responsive stimulation for the long term.
  Interventions: Device: RNS System

INTERVENTIONS:
Device: RNS System — The RNS System provides closed loop responsive brain stimulation. In response to detection of previously identified electrocorticographic activity, the neurostimulator delivers stimulation to the seizure foci by way of the leads to interrupt the activity before the patient experiences clinical seizures. The typical patient is treated with a cumulative total of 5 minutes of stimulation a day.

SUMMARY:
The purpose of the study is to follow patients with partial onset seizures prospectively over 5 years in the real-world environment to gather data on the long-term safety and effectiveness of the RNS System at qualified CECs by qualified neurologists, epileptologists, and neurosurgeons trained on the RNS System.

DETAILED DESCRIPTION:
NeuroPace, Inc. is sponsoring a post-approval study (PAS) of the RNS System device. The RNS System is the first FDA-approved closed loop responsive neurostimulator designed to reduce the frequency of seizures in individuals with partial onset seizures.

The RNS System Epilepsy PAS is a 5 year, non-randomized, open-label, multi-center prospective observational study. Data regarding safety and efficacy are collected at enrollment and periodically throughout the 5-year study.

The study is designed to assess the long-term safety and effectiveness of the RNS System as an adjunctive therapy in reducing the frequency of seizures in individuals 18 years of age or older with partial onset seizures who have undergone diagnostic testing that localized no more than 2 epileptogenic foci, are refractory to two or more antiepileptic medications, and currently have frequent and disabling seizures (motor partial seizures, complex partial seizures and/or secondarily generalized seizures).

Data from the RNS System Epilepsy PAS will be used to calculate long-term SAE rates, median percent change in seizure frequency (from pre-implant retrospective data), as well as other safety and effectiveness endpoints.

ELIGIBILITY:
Inclusion Criteria:

A clinical decision to treat the patient with the RNS System in accordance with its approved indication for use has been made prior to enrollment in the study. For approved indication for use and contraindications, refer to current physician labeling and instructions for use (manuals) for the RNS System available at the NeuroPace website (www.neuropace.com).

This post-approval study also has the following additional study related inclusion criteria:

* Subject or legal guardian is able to provide appropriate consent to participate
* Subject is able to maintain a seizure diary alone or with the assistance of a competent individual
* Subject is able to attend clinic appointments in accordance with the study schedule

Exclusion Criteria:

Per clinician assessment, treatment with the RNS System is contraindicated based on current RNS System labeling. For approved indication for use and contraindications, refer to current physician labeling and instructions for use (manuals) for the RNS System available at the NeuroPace website (www.neuropace.com).

This post-approval study has the following additional study related exclusion criteria:

* Subject is participating in a therapeutic investigational drug or device study
* Subject was treated with a VNS within the last three months (90 days)
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years of age or older with partial onset seizures who have undergone diagnostic testing that localized no more than 2 epileptogenic foci, are refractory to two or more antiepileptic medications, and currently have frequent and disabling seizures.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
SAE rate | Implant through 5 years post-implant
  Calculate annual SAE rates over time in the entire subject population as well as within subpopulations.
Neurosurgeon experience | Implant through 41 days post-implant
  Demonstrate there is no difference in safety in 6-week perioperative period based on the experience of NeuroPace qualified and trained implanting physicians.
Physician experience | Implant through 1 year post-implant
  Demonstrate there is no difference in safety 1 year post-implant based on experience of NeuroPace qualified and trained treating physicians and Comprehensive Epilepsy Centers.
Product use - surgical procedures
  Present the incidence and number of AEs related to surgical procedures associated with implant, explant, reimplantation, and revision of the neurostimulator and lead(s).
Autopsy
  Present data from autopsies obtained from any patient implanted with neurostimulator/leads.
Median percentage reduction in disabling seizure | Pre-implant (retrospective data) compared to 30 to 36 months post-implant
  Demonstrate that the median percentage reduction in disabling seizures over time in the entire subject population is comparable to the median percentage reduction in disabling seizures over time in the LTT study. Characterize the median percentage reduction in disabling seizures over time within subpopulations.
Neurostimulator programming | Through 5 years post-implant
  Demonstrate that stimulation programming classes have similar effects on the overall seizure frequency.

SECONDARY OUTCOMES:
Seizure worsening | 6 months post-implant through 36 months post-implant
  Demonstrate that there is not a worsening in disabling seizures over time in the entire subject population. Assess the sustained effect on disabling seizure frequency over time within subpopulations.
Neurostimulator programming | Implant through 5 years post-implant
  Characterize the effects of stimulation programming classes on the overall 5-year rate of SAEs and device-related non-serious AEs.

OTHER OUTCOMES:
Neurostimulator battery longevity
  Characterize the clinically observed battery longevity over time and in relation to therapy load in patients treated with the RNS System.

CONTACTS AND LOCATIONS:
Overall Officials: Martha J Morrell, MD, Study Director — NeuroPace, Inc.
Locations (35):
- United States (35):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Cente, Lebanon, New Hampshire
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Pennsylvania State University / Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Seton Family of Hospital, Austin, Texas
  - Austin Epilepsy Care Center, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Intermountain Healthcare Research, Salt Lake City, Utah
  - University of Washington Harborview Medical Center, Seattle, Washington
  - Swedish Health Services, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergey GK, Morrell MJ, Mizrahi EM, Goldman A, King-Stephens D, Nair D, Srinivasan S, Jobst B, Gross RE, Shields DC, Barkley G, Salanova V, Olejniczak P, Cole A, Cash SS, Noe K, Wharen R, Worrell G, Murro AM, Edwards J, Duchowny M, Spencer D, Smith M, Geller E, Gwinn R, Skidmore C, Eisenschenk S, Berg M, Heck C, Van Ness P, Fountain N, Rutecki P, Massey A, O'Donovan C, Labar D, Duckrow RB, Hirsch LJ, Courtney T, Sun FT, Seale CG. Long-term treatment with responsive brain stimulation in adults with refractory partial seizures. Neurology. 2015 Feb 24;84(8):810-7. doi: 10.1212/WNL.0000000000001280. Epub 2015 Jan 23. PMID 25616485
- [Background] Heck CN, King-Stephens D, Massey AD, Nair DR, Jobst BC, Barkley GL, Salanova V, Cole AJ, Smith MC, Gwinn RP, Skidmore C, Van Ness PC, Bergey GK, Park YD, Miller I, Geller E, Rutecki PA, Zimmerman R, Spencer DC, Goldman A, Edwards JC, Leiphart JW, Wharen RE, Fessler J, Fountain NB, Worrell GA, Gross RE, Eisenschenk S, Duckrow RB, Hirsch LJ, Bazil C, O'Donovan CA, Sun FT, Courtney TA, Seale CG, Morrell MJ. Two-year seizure reduction in adults with medically intractable partial onset epilepsy treated with responsive neurostimulation: final results of the RNS System Pivotal trial. Epilepsia. 2014 Mar;55(3):432-41. doi: 10.1111/epi.12534. Epub 2014 Feb 22. PMID 24621228
- [Background] Morrell MJ; RNS System in Epilepsy Study Group. Responsive cortical stimulation for the treatment of medically intractable partial epilepsy. Neurology. 2011 Sep 27;77(13):1295-304. doi: 10.1212/WNL.0b013e3182302056. Epub 2011 Sep 14. PMID 21917777